CLINICAL TRIAL: NCT01107405
Title: Efficacy of Loteprednol Etabonate Ophthalmic Base Compared to Loteprednol Etabonate Ophthalmic Suspension vs Placebo in a Modified Conjunctival Allergen Challenge(CAC) Model
Brief Title: Loteprednol Ophthalmic Base Compared to Loteprednol Ophthalmic Suspension vs Placebo in an Allergen Challenge
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 584
Record Dates: First submitted 2010-04-15; First posted 2010-04-21 (Estimated); Results first posted 2012-03-21 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-02

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — BID protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Loteprednol etabonate base (QD) (Active Comparator): Loteprednol etabonate ophthalmic base dosed once/day.
  Interventions: Drug: Loteprednol etabonate base (QD)
- Loteprednol etabonate base (BID) (Active Comparator): Loteprednol etabonate ophthalmic base dosed two times/day
  Interventions: Drug: Loteprednol etabonate base (BID)
- Loteprednol etabonate base (QID) (Active Comparator): Loteprednol etabonate ophthalmic base dosed four times/day.
  Interventions: Drug: Loteprednol etabonate base (QID)
- Loteprednol etabonate suspension (QID) (Active Comparator): Loteprednol etabonate ophthalmic suspension dosed four times/day
  Interventions: Drug: Loteprednol etabonate suspension
- Vehicle of loteprednol etabonate (Placebo Comparator): Vehicle of loteprednol etabonate, dosed either QD, BID, or QID
  Interventions: Drug: Vehicle of loteprednol etabonate

INTERVENTIONS:
Drug: Loteprednol etabonate base (QD) — Loteprednol Etabonate ophthalmic base once daily dosing for 2 weeks
  Arms: Loteprednol etabonate base (QD)
Drug: Loteprednol etabonate base (BID) — Loteprednol etabonate ophthalmic base BID dosing for 2 weeks
  Arms: Loteprednol etabonate base (BID)
Drug: Loteprednol etabonate base (QID) — Loteprednol Etabonate ophthalmic base four times/day dosing for 2 week
  Arms: Loteprednol etabonate base (QID)
Drug: Loteprednol etabonate suspension — Loteprednol etabonate ophthalmic suspension dosed four times daily for 2 weeks.
  Arms: Loteprednol etabonate suspension (QID)
Drug: Vehicle of loteprednol etabonate — Vehicle of loteprednol etabonate ophthalmic dosed once, twice or four times daily for 2 weeks.
  Arms: Vehicle of loteprednol etabonate

SUMMARY:
The purpose of this study is to evaluate the efficacy of loteprednol etabonate ophthalmic base, compared to loteprednol etabonate ophthalmic suspension, and vehicle in the prevention of the signs and symptoms of allergic conjunctivitis in a modified Conjunctival Allergen Challenge model and in an environmental model during pollen season. Comparisons will be made following 2 weeks of dosing.

ELIGIBILITY:
Inclusion Criteria:

* Positive history of ocular allergies and positive skin test reaction to cat hair, cat dander, grasses, ragweed, and/or trees within the past 24 months.
* Calculated best-corrected visual acuity of 0.70 logMAR or better in each eye as measured using the ETDRS chart.
* Positive bilateral conjunctival allergen challenge(CAC)reaction within 10 minutes of instillation of the last titration of allergen at visit 1.
* Positive bilateral CAC reaction in 1 out of 3 time points for the initial and re-challenge at visit 2.

Exclusion Criteria:

* Known contraindications or sensitivities to the study medication or its components.
* Any ocular condition that, in the opinion of the investigator, could affect the subjects safety or trial parameters.
* Use of disallowed medications during the period indicated prior to study enrollment or during the study.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2010-04; Primary Completion 2010-05 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tuyen Ong, MD, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This 2 week ocular allergy study was conducted at 2 ophthalmology clinics in the United States. The first participant was enrolled on 4/22/2010 and the last participant visit was 5/30/2010.
Pre-assignment Details: 238 participants were screened, a total of 101 participants with seasonal and perennial allergy were randomized into the study. These 101 participants comprised the safety population, 90 of which completed the study. The ITT population was comprised of 97 subjects (4 excluded due to no post CAC-assessment).
Period: Overall Study
Arm/Group | Loteprednol Etabonate Base (QD) | Loteprednol Etabonate Base (BID) | Loteprednol Etabonate Base (QID) | Loteprednol Etabonate Suspension (QID) | Vehicle of Loteprednol Etabonate
Started | 21 | 20 | 20 | 20 | 20
Completed | 19 | 19 | 18 | 17 | 17
Not Completed | 2 | 1 | 2 | 3 | 3
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 2 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Loteprednol Etabonate Base (QD) | Loteprednol Etabonate Base (BID) | Loteprednol Etabonate Base (QID) | Loteprednol Etabonate Suspension (QID) | Vehicle of Loteprednol Etabonate | Total
Number analyzed (Participants) | 21 | 20 | 20 | 20 | 20 | 101
Age, Customized [Number; unit: participants]
  <=19 years | 3 | 1 | 1 | 1 | 2 | 8
  20 - 64 years | 18 | 18 | 18 | 19 | 18 | 91
  >=65 years | 0 | 1 | 1 | 0 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 13 | 9 | 12 | 60
  Male | 8 | 7 | 7 | 11 | 8 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 1 | 0 | 3
  Not Hispanic or Latino | 19 | 20 | 20 | 19 | 20 | 98
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching
Description: Evaluated by subject at 3, 5, and 7 min post challenge on a scale of 0-4 where 0=no itching and 4=incapacitating itch.
Time Frame: Visit 4 (8 hr re-challenge)
Population: Visit 4, Re-challenge Ocular Itching Scores - Primary Analysis ITT Population with LOCF included data from all randomized subjects who received treatment and had at least 1 post-CAC assessment.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Loteprednol Etabonate Base (QD) | Loteprednol Etabonate Base (BID) | Loteprednol Etabonate Base (QID) | Loteprednol Etabonate Suspension (QID) | Vehicle of Loteprednol Etabonate
Number analyzed (Participants) | 21 | 20 | 18 | 19 | 19
Units on a Scale
  3 Min | 1.48 (1.040) | 1.84 (0.978) | 1.82 (0.954) | 1.93 (0.794) | 2.68 (0.916)
  5 Min | 1.63 (1.036) | 2.13 (0.988) | 1.96 (0.960) | 2.12 (0.918) | 2.78 (0.924)
  7 Min | 1.54 (1.035) | 2.03 (1.097) | 1.89 (0.993) | 2.04 (0.951) | 2.71 (0.899)

2. Primary Outcome: Conjunctival Redness
Description: Evaluated by investigator at 7, 15 and 20 minutes post challenge on a scale of 0-4 where 0= no redness and 4=extremely severe redness.
Time Frame: Visit 4 (8 hr re-challenge)
Population: Visit 4, Re-challenge Conjunctival Hyperemia Scores, ITT Population with LOCF included data from all randomized subjects who received treatment and had at least 1 post-CAC assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Loteprednol Etabonate Base (QD) | Loteprednol Etabonate Base (BID) | Loteprednol Etabonate Base (QID) | Loteprednol Etabonate Suspension (QID) | Vehicle of Loteprednol Etabonate
Number analyzed (Participants) | 21 | 20 | 18 | 19 | 19
Units on a scale
  7 min | 1.76 (0.620) | 1.99 (0.709) | 2.11 (0.649) | 2.16 (0.619) | 2.59 (0.501)
  15 min | 1.95 (0.660) | 2.13 (0.829) | 2.28 (0.766) | 2.18 (0.600) | 2.71 (0.597)
  20 min | 2.02 (0.720) | 2.06 (0.811) | 2.28 (0.691) | 2.16 (0.585) | 2.74 (0.592)

3. Secondary Outcome: Ocular Itching
Description: Evaluated by the subject at 3, 5 and 7 min post-challenge on a scale of 0-4 where 0=no itching and 4=incapacitating itch.
Time Frame: Visit 3 (initial challenge)
Population: Visit 3 Ocular Itching Scores - ITT Population with LOCF included data from all randomized subjects who received treatment and had at least 1 post-CAC assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Loteprednol Etabonate Base (QD) | Loteprednol Etabonate Base (BID) | Loteprednol Etabonate Base (QID) | Loteprednol Etabonate Suspension (QID) | Vehicle of Loteprednol Etabonate
Number analyzed (Participants) | 21 | 20 | 18 | 19 | 19
units on a scale
  3 Min | 2.50 (0.829) | 2.00 (0.778) | 2.31 (0.889) | 2.28 (0.946) | 2.50 (1.000)
  5 min | 2.45 (0.781) | 2.15 (0.745) | 2.46 (1.016) | 2.47 (0.979) | 2.63 (0.863)
  7 min | 2.38 (0.872) | 2.21 (0.783) | 2.21 (1.044) | 2.38 (1.062) | 2.45 (0.810)

4. Secondary Outcome: Conjunctival Redness
Description: as for outcome 2
Time Frame: Visit 3 (initial challenge)
Population: Visit 3 Conjunctival Hyperemia Scores - ITT Population with LOCF included data from all randomized subjects who received treatment and had at least 1 post-CAC assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Loteprednol Etabonate Base (QD) | Loteprednol Etabonate Base (BID) | Loteprednol Etabonate Base (QID) | Loteprednol Etabonate Suspension (QID) | Vehicle of Loteprednol Etabonate
Number analyzed (Participants) | 21 | 20 | 18 | 19 | 19
units on a scale
  7 min | 2.14 (0.584) | 2.05 (0.484) | 2.22 (0.593) | 2.25 (0.486) | 2.41 (0.663)
  15 min | 2.26 (0.509) | 2.20 (0.737) | 2.28 (0.664) | 2.43 (0.415) | 2.42 (0.795)
  20 min | 2.31 (0.541) | 2.24 (0.631) | 2.18 (0.706) | 2.33 (0.590) | 2.42 (0.834)

5. Secondary Outcome: Ocular Itching
Description: as for outcome 3
Time Frame: Visit 4 (initial challenge)
Population: Visit 4 Ocular Itching Scores - ITT Population with LOCF included data from all randomized subjects who received treatment and had at least 1 post-CAC assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Loteprednol Etabonate Base (QD) | Loteprednol Etabonate Base (BID) | Loteprednol Etabonate Base (QID) | Loteprednol Etabonate Suspension (QID) | Vehicle of Loteprednol Etabonate
Number analyzed (Participants) | 21 | 20 | 18 | 19 | 19
units on a scale
  3 Min | 2.02 (0.978) | 1.93 (1.130) | 2.04 (0.913) | 2.17 (0.846) | 2.55 (0.880)
  5 min | 2.19 (1.040) | 2.14 (1.071) | 2.15 (0.888) | 2.32 (0.853) | 2.82 (0.877)
  7 min | 2.11 (1.026) | 2.11 (0.985) | 2.13 (0.917) | 2.22 (0.953) | 2.71 (0.875)

6. Secondary Outcome: Conjunctival Redness
Description: as for outcome 2
Time Frame: Visit 4 (initial challenge)
Population: Visit 4 Conjunctival Hyperemia Scores - ITT Population with LOCF included data from all randomized subjects who received treatment and had at least 1 post-CAC assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Loteprednol Etabonate Base (QD) | Loteprednol Etabonate Base (BID) | Loteprednol Etabonate Base (QID) | Loteprednol Etabonate Suspension (QID) | Vehicle of Loteprednol Etabonate
Number analyzed (Participants) | 21 | 20 | 18 | 19 | 19
units on a scale
  7 min | 1.96 (0.755) | 2.19 (0.683) | 2.26 (0.661) | 2.22 (0.353) | 2.70 (0.445)
  15 min | 2.05 (0.793) | 2.19 (0.777) | 2.28 (0.717) | 2.36 (0.459) | 2.83 (0.479)
  20 min | 2.15 (0.777) | 2.16 (0.828) | 2.28 (0.701) | 2.29 (0.573) | 2.80 (0.544)

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Loteprednol Etabonate Base (QD) | Loteprednol Etabonate Base (BID) | Loteprednol Etabonate Base (QID) | Loteprednol Etabonate Suspension (QID) | Vehicle of Loteprednol Etabonate
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/21 | 4/20 | 5/20 | 1/20 | 6/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Loteprednol Etabonate Base (QD) (N=21) | Loteprednol Etabonate Base (BID) (N=20) | Loteprednol Etabonate Base (QID) (N=20) | Loteprednol Etabonate Suspension (QID) (N=20) | Vehicle of Loteprednol Etabonate (N=20)
Eye irritation (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (2)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pruritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngial pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post nasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood oestrogen decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to any presentation of results, draft versions of manuscripts will be made available to co-authors and to the Sponsor for review and comment. At least 30 days in the case of abstracts or 60 days in the case of full papers should be allowed for comments prior to submission for consideration of acceptance of presentation or publication.